CLINICAL TRIAL: NCT01441128
Title: A Phase 1, Open-Label, Dose Escalation Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of Combined Oral C-Met/ALK Inhibitor (PF-02341066) and Pan-Her Inhibitor (PF-0299804) in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: -02341066 and PF-00299804 for Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110250; 11-C-0250
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-02-26

CONDITIONS: Carcinoma, Non-Small Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell; Carcinoma, Large Cell
Keywords: Lung Neoplasms; Epithelial-Mesenchymal Transition Factor (c-Met); Tyrosine Kinase Inhibitor; Hepatocyte Growth Factor Receptor; Epidermal Growth Factor Receptor; Non Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma, Squamous Cell; Carcinoma, Large Cell; Lung Neoplasms

ARMS (2):
- Arm 1 (Experimental): The starting doses will be 200 mg by mouth, twice a day of PF 02341066 in tablet form and 30 mg by mouth once a day of PF 0029804 in tablet form. Thedose of each drug in the combination will be escalated or de-escalated until the maximum tolerated combined dose is reached. Patients will then be treated with the maximum tolerated combined dose.
  Interventions: Drug: PF-02341066/PF-00299804
- Arm 2 (Experimental): 45 mg by mouth once a day of PF-00299804 in tablet form until progressive disease and then the maximum tolerated combined dose of PF-02341066 (given by mouth twice a day in tablet form) and PF-00299804 (given by mouth once a day in tablet form).
  Interventions: Drug: PF-02341066/PF-00299804

INTERVENTIONS:
Drug: PF-02341066/PF-00299804 — Combined PF-02341066 and PF-00299804
Drug: PF-02341066/PF-00299804 — Single Agent PF-00299804 followed by Combined PF-02341066 and PF-00299804

SUMMARY:
Background:

- PF-02341066 and PF-00299804 are drugs that specifically target certain proteins that may be more active in cancer cells than normal cells, in particular in non-small cell lung cancer. Both drugs seem to be able to stop the growth of or kill cancer cells. Researchers want to combine them to see if they are a safe and effective treatment for advanced non-small cell lung cancer.

Objectives:

- To test the safety and effectiveness of PF-02341066 and PF-00299804 for advanced non-small cell lung cancer.

Eligibility:

- Individuals at least 18 years of age with advanced non-small cell lung cancer that has not responded to standard treatments.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood and urine tests, and imaging studies. Heart and lung function tests and an eye exam may also be given.
* The first cycle of treatment will be 28 days. Every cycle after the first will be 21 days. Participants may have up to 17 cycles of treatment.
* Participants will take both study drugs as tablets. Twelve hours after the first dose, participants will take only the PF-02341066. This dose schedule will remain the same throughout the study.
* Participants will be monitored with frequent blood and urine tests and imaging studies. Tumor biopsies will be taken as needed. Those in the study will keep a diary to record any symptoms or side effects of taking the study drugs.
* After 17 cycles of treatment, or after stopping the study drugs early for any other reason, participants will have a final followup visit.

DETAILED DESCRIPTION:
BACKGROUND:

* Approximately 85% of lung cancer is defined histologically as NSCLC and the majority of patients present with inoperable locally advanced (Stage IIIB) or metastatic (Stage IV) disease for which no curative treatment is available.
* Patients with disease progression on or after first-line treatment with platinum-based doublets may be candidates for second-line treatment.
* Recent evidence strongly implicates EGFR activating somatic mutations as a mechanism of tumorigenesis and a determinant of sensitivity to EGFR TKIs in NSCLC.
* Despite the dramatic initial response to gefitinib and erlotinib, about 50% of NSCLC tumors develop resistance due to secondary activating mutations in EGFR itself, including the EGFR T790M gatekeeper mutation, and more than 20% of acquired resistance is due to an increase in mesenchymal-epithelial transition factor (c-Met) signaling.
* There is evidence from a limited number of tumors from patients with acquired resistance to EGFR-TKIs that both T790M and cMET resistance mechanisms can occur in the same patient at different metastatic sites and even in different fractions of the same lesion.
* Tumors with acquired resistance to erlotinib and gefitinib might be vulnerable to a combination of PF-00299804 a second generation EGFR TKI which is also an inhibitor of T790M mutation, and PF-02341066 which is an inhibitor of c- Met/Hepatocyte Growth Factor Receptor (HGFR).

OBJECTIVES:

- To define the recommended Phase 2 dose (RP2D) of combined PF-02341066 plus

PF-00299804 in patients with advanced Non-Small Cell Lung Cancer (NSCLC).

* To assess the overall safety and tolerability, plasma pharmacokinetics (PK) and clinical activity of combined PF-02341066 plus PF-00299804.
* To analyze potential predictive and pharmacodynamic biomarkers in tumor and blood in patients with advanced NSCLC who have acquired resistance to erlotinib or gefitinib

ELIGIBILITY:

* Dose Escalation Phase: Adults with histologically documented diagnosis of NSCLC that is locally advanced or metastatic, after failure of either at least one chemotherapy regimen or treatment with erlotinib or gefitinib.
* Expansion Phase: Adults with histologically documented diagnosis of NSCLC that is locally advanced or metastatic, with acquired resistance to erlotinib or gefitinib, and must have one lesion amendable to biopsy.
* All pathology samples will be reviewed at the NCI.

DESIGN:

* Phase 1, multi-center, open-label, non-randomized trial of combined oral PF- 02341066 and oral PF-00299804 in patients with advanced NSCLC. Trial consists of two phases.
* Dose Escalation Phase: Patients will be treated with varying doses of combined PF- 02341066 plus PF-00299804. Tumor biopsy is not required.
* Expansion Phase: Two expansion cohorts will run concurrently following completion of the Dose Escalation Phase. Both cohorts will enroll patients with locally advanced or metastatic NSCLC with acquired resistance to erlotinib or gefitinib, which is defined as progression following an initial response (complete or partial) or stable disease for at least six months while on erlotinib or gefitinib.
* The dose escalation phase and the dose expansion phase can run concurrently insofar as the dose expansion phase can enroll before completion of the dose escalation phase provided that the dose used in the expansion phase has already been tested in the escalation phase and has been declared safe; i.e., for each specific safe dose the escalation phase is followed by the expansion phase.
* Tumor biopsy is mandatory for Expansion Phase entrance, however, all patients will be treated with study drugs irrespective of the biomarker identified which will be analyzed retrospectively. The mandatory biopsy in the Expansion Phase is necessary in order to identify acquired mutations that change over time.
* Expansion cohort 1 will continue to evaluate safety, tolerability and PK of the drug combination PF-02341066 plus PF-00299804.
* Expansion cohort 2 will enroll patients who are either untreated by prior PF- 00299804 or who have progressed on single agent PF-00299804 administered in an ongoing clinical trial. Patients who are previously untreated with PF-00299804 will be treated sequentially; i.e., first with single agent PF-00299804 until progression, then with the combination of PF-02341066 plus PF-00299804. Those who progressed with single agent PF-00299804 on another clinical trial will be treated with the combination PF-02341066 plus PF-00299804.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject eligibility should be reviewed and documented by an appropriately qualified member of the investigator s study team before subjects are included in the study.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:
* Disease Criteria:
* Dose Escalation Phase: Histologically proven diagnosis of NSCLC that is locally advanced or metastatic, after failure of either at least one prior chemotherapy regimen or targeted therapy.
* Expansion Phase: Histologically proven diagnosis of NSCLC that is locally advanced or metastatic and with acquired resistance to erlotinib or gefitinib. Acquired resistance is defined as progression following either an initial response (complete or partial), or stable disease for at least six months, while on single agent erlotinib or single agent gefitinib. In addition to these patients, Cohort 2 will also enroll patients from ongoing trials, including A7471017 and A7471028, who have progressed on single agent PF-00299804.
* For the dose escalation phase, any prior treatment (chemotherapy, targeted therapy, radiation or surgery) must have been completed at least 2 weeks prior to initiation of study medication, except patients being treated with single agent PF-02341066 will have the option of continuing single agent PF-02341066 until the combination of PF- 02341066 and PF-00299804 is given. For the expansion phase, patients must not have had any intervening treatmen (chemotherapy, targeted therapy, radiation or surgery) between single agent erlotinib or single agent gefitinib treatment, and biopsy and dosing with study drug, unless agreed by the sponsor. In Expansion Cohort 2, patients who have received PF-00299804 as part of an ongoing clinical trial will continue with single agent therapy with PF-00299804 at their current dose after documentation of progression until the combination is given.
* Any acute toxicity from prior treatment must have been recovered to less than or equal to Grade 1 (except alopecia).
* At least 1 target lesion used for assessment of antitumor activity must be measurable by RECIST (version 1.1), or considered evaluable by agreement between the investigator and the sponsor.
* Target lesions can be chosen from a previous irradiated area if lesions in those areas have documented progression.
* Female or male, 18 years of age or older.
* ECOG (Zubrod) performance status 0-2.
* Adequate organ function as defined by the following criteria measured within 7 days prior to enrollment.
* Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) less than or equal to 2.5 times upper limit of normal (ULN), or AST and ALT less than or equal to 5 times ULN if liver function abnormalities are due to underlying malignancy;
* Total serum bilirubin less than or equal to 1.5 times ULN (except patients with documented Gilbert s syndrome);
* Absolute neutrophil count (ANC) greater than or equal to1000/microL;
* Platelets greater than or equal to 30,000/microL;
* Hemoglobin greater than or equal to 8.0 g/dl;
* Serum creatinine <2 times institution ULN.
* Adequate cardiac function, including:
* 12-Lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention;
* QTc interval less than or equal to 470 msec and without history of Torsades de Pointes or other symptomatic QTc abnormality;
* LVEF (by MUGA or echocardiogram) of greater than or equal to 50%.
* All female patients of child-bearing potential are required to have a negative pregnancy test at screening. The test should be repeated whenever one menstrual cycle is missed during treatment or a potential pregnancy is otherwise suspected.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, other study procedures and, for enrollment into the Expansion Phase, must be willing to undergo a tumor biopsy.

EXCLUSION CRITERIA:

Subjects presenting with any of the following will not be included in the study:

* Participation in other studies or treatment within 2 weeks before the current study begins and/or during study participation (with the exception of patients who are receiving single agent PF-00299804 and who enroll into Expansion Cohort 2 from ongoing trials including A7471017 and A7471028, and with the exception of patients being treated with single agent PF-02341066 treatment who enroll during the dose escalation phase and exercise the option of continuing single agent PF-02341066 treatment until the combination of PF-02341066 and PF-00299804 is given) to allow for recovery and drug wash-out.
* Known interstitial fibrosis or interstitial lung disease.
* Patients with known brain metastases who are neurologically stable (asymptomatic) for at least 2 weeks and with no ongoing requirement for corticosteroids may enroll on study before treatment of brain metastases.
* History of carcinomatous meningitis, or leptomeningeal disease.
* Any of the following within 6 months prior to starting study treatment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack.
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation or Torsades de Pointes). Diagnosed or suspected congenital long QT syndrome. Ongoing cardiac dysrhythmias of Grade greater than or equal to 2 (CTCAE version 4.02), uncontrolled atrial fibrillation of any grade, or QTc interval >470 msec.
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
* Patient must not have had major surgery or trauma within 28 days prior to enrollment.
* Active uncontrolled infection.
* Pregnant or lactating females.
* Significant gastrointestinal condition that may impair intake, transit, absorption or ability to tolerate investigational drugs.
* Prior malignancy (other than NSCLC): patients will not be eligible if they have evidence of active malignancy (other than non-melanoma skin cancer or in situ cervical cancer, or localized and presumed cured prostate cancer with PSA < ULN) within the last 3 years.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Use of drugs or foods that are known potent CYP3A4 inhibitors within 7 days prior to the first dose of study medication, including but not limited to itraconazole, ketoconazole, miconazole, clarithromycin, erythromycin, indinavir, nefazodone, amprenavir, delavirdine, nelfinavir, ritonavir, saquinavir, diltiazem, verapamil and grapefruit juice.
* Use of drugs that are known potent CYP3A4 inducers within 12 days prior to the first dose of study medication, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifabutin, rifampin, tipranavir, ritonavir, and St. John s wort.
* Concurrent use of drugs that are CYP3A4 substrates with narrow therapeutic indices, including but not limited to pimozide, aripiprazole, triazolam, ergotamine and halofantrine.
* Concurrent use of drug that are highly dependent on CYP2D6 metabolism including S-metoprolol, propafenone, timolol, amitriptyline, clomipramine, desipramine, imipramine, paroxetine, haloperidol, risperidone, thioridazine, codeine, flecainide, mexilletine, tamoxifen, venlafaxine.

Dextromethorphan, a CYP2D6, substrate is allowed if medically indicated and no suitable alternative anti-tussive medication is available. However, the dose of dextromethorphan may need to be modified. In a clinical study in healthy volunteers who were extensive metabolizers (A7471039) PF-00299804 increased mean total exposure (AUC(last) and C(max)) of dextromethorphan 855% and 874%, respectively, following concomitant administration with PF-00299804 45 mg compared to exposure of administration of dextromethorphan alone. Extensive metabolizers comprise approximately 80% of the population, with ultra-, intermediate-, and poor-metabolizers accounting for the remaining portion of the general population. Therefore, if no alternative is available dextromethorphan dosing should be initiated at a lower dose (approx 25%) with close monitoring of patient clinical status. Dose increases or decreases of dextromethorphan may be considered based upon individual patient tolerability.

Lidocaine may be used systemically with clinical monitoring (including telemetry).

Opiates such as morphine, oxycodone, dihydrocodeine, hydrocodone, and tramadol can be used as substitutes to replace codeine. Use of these opiates should be monitored for altered analgesic effect during treatment as they may be partly metabolized by CYP2D6.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09-01; Primary Completion 2014-02-28 (Actual); Study Completion 2015-02-26 (Actual)

PRIMARY OUTCOMES:
Overall safety profile of combined PF 02341066 plus PF 00299804 including adverse events (AE), as defined and graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], and first cycle Dose Limiting Tox... | 18 months

SECONDARY OUTCOMES:
Plasma concentrations and pharmacokinetic (PK) parameters of PF 02341066 and PF 00299804 including AUCtau, Cmax, Ctrough, Tmax, and CLss/F | 18 months
Clinical activity of combined PF 02341066 plus PF 00299804 including objective response (OR) and stable disease (SD) as defined by RECIST version 1.1, duration of response (DR) and progression free survival (PFS). | 18 months
Biomarkers in tumor and blood that are potentially predictive for drug activity: for example, KRAS mutations, EGFR mutations (eg, T790M), EGFR and HER2 amplifications, c Met amplification and mutations, ALK, PTEN and PIK3A status in tumor biopsi... | 12 months
Pharmacodynamic biomarkers in tumor biopsies (e.g., phospho c Met, c Met, EGFR, phospho EGFR) and in blood (e.g., HGF and s Met) that are modulated following drug exposure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alberola V, Camps C, Provencio M, Isla D, Rosell R, Vadell C, Bover I, Ruiz-Casado A, Azagra P, Jimenez U, Gonzalez-Larriba JL, Diz P, Cardenal F, Artal A, Carrato A, Morales S, Sanchez JJ, de las Penas R, Felip E, Lopez-Vivanco G; Spanish Lung Cancer Group. Cisplatin plus gemcitabine versus a cisplatin-based triplet versus nonplatinum sequential doublets in advanced non-small-cell lung cancer: a Spanish Lung Cancer Group phase III randomized trial. J Clin Oncol. 2003 Sep 1;21(17):3207-13. doi: 10.1200/JCO.2003.12.038. PMID 12947054
- [Background] Kelly K, Crowley J, Bunn PA Jr, Presant CA, Grevstad PK, Moinpour CM, Ramsey SD, Wozniak AJ, Weiss GR, Moore DF, Israel VK, Livingston RB, Gandara DR. Randomized phase III trial of paclitaxel plus carboplatin versus vinorelbine plus cisplatin in the treatment of patients with advanced non--small-cell lung cancer: a Southwest Oncology Group trial. J Clin Oncol. 2001 Jul 1;19(13):3210-8. doi: 10.1200/JCO.2001.19.13.3210. PMID 11432888
- [Background] Scagliotti GV, De Marinis F, Rinaldi M, Crino L, Gridelli C, Ricci S, Matano E, Boni C, Marangolo M, Failla G, Altavilla G, Adamo V, Ceribelli A, Clerici M, Di Costanzo F, Frontini L, Tonato M; Italian Lung Cancer Project. Phase III randomized trial comparing three platinum-based doublets in advanced non-small-cell lung cancer. J Clin Oncol. 2002 Nov 1;20(21):4285-91. doi: 10.1200/JCO.2002.02.068. PMID 12409326